CLINICAL TRIAL: NCT00826761
Title: Probiotics and Satiety - Acute Effects and Persistence of Acute Effects
Brief Title: ProSat - Effect of Probiotics on Satiety
Acronym: ProSat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Chr Hansen A/S (Unknown)
Responsible Party: Principal Investigator, AAstrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B257
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Appetite Regulation
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Active Comparator): High dose Lb. casei
  Interventions: Dietary Supplement: probiotic
- 2 (Active Comparator): Low dose Lb. Casei
  Interventions: Dietary Supplement: probiotic
- 3 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotic — One capsule per meal test (high dose or low dose)
  Arms: 1; 2
Dietary Supplement: placebo — 1 capsuel every morning
  Arms: 3

SUMMARY:
The aim of the ProSat study is to examine the effects of a probiotic capsule containing one of two doses (low and high dose) of Lb. Casei on subjective appetite sensation, ad libitum energy intake, and appetite hormone response in a single meal test and to determine whether the acute effects persist after daily supplementation of the probiotic capsule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Normal to slight overweight (BMI: 22-28 kg/m2)
* 20-45 years of age

Exclusion Criteria:

* Smoking
* Daily medicine use (oral contraceptives excluded)
* Use of pre- and probiotic supplements and foods
* Blood donation 3 months prior to the study
* Hb<8mmol/l
* Chronic illnesses such as hyperlipidemia, diabetes inflammatory diseases
* Pregnancy or breastfeeding
* Elite athletes (>10 hours hard exercise/week)
* Vegetarians

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Glucose; Insulin; GLP-1; CCK; PYY; grehlin; PP; amylin; LPS; TNF-alfa; hsCRP; fibrinogen | 2013

SECONDARY OUTCOMES:
Subjective appetite measurements; Spontaneous food intake | 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark